CLINICAL TRIAL: NCT03817203
Title: Assistant Professor, Physioterapist, PhD
Brief Title: Effects of Kinesio Taping Application in Women With Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, Assistant Professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/08/05
Record Dates: First submitted 2019-01-20; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio tape group (Experimental): Kinesio tape application and pelvic floor exercise have been applied
  Interventions: Other: Kinesio tape application
- Control group (Sham Comparator): Sham kinesio tape application and pelvic floor exercise have been applied
  Interventions: Other: Sham tape application

INTERVENTIONS:
Other: Kinesio tape application — Kinesio tape application combined with pelvic floor exercises will be performed.Taping is carried out for 2 days/week in 6 weeks. The exercise program is performed every day for 6 weeks
  Arms: Kinesio tape group
Other: Sham tape application — Sham tape application combined with pelvic floor exercises will be performed.Sham taping is carried out for 2 days/week in 6 weeks. The exercise program is performed every day for 6 weeks
  Arms: Control group

SUMMARY:
The aim of this study is to compare the effects of kinesio tape application on bladder symptoms and quality of life in women with overactive bladder (OAB).

ELIGIBILITY:
Inclusion Criteria:

* 20 to 65 years of age,
* having overactive bladder
* being volunteer

Exclusion Criteria:

* pregnancy,
* only stress incontinence,
* the presence of a malignant condition with a history of acute infection,
* having a mental problem to prevent co-morbidity, evaluation and cooperative

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
The severity of overactive bladder symptoms assessed with Overactive Bladder Questionnaire_V8 | Change from baseline bladder symptoms at 6 weeks
  Overactive Bladder Questionnaire_V8 assessing severity of overactive bladder symptoms will be used. This scale includes items on urgency, incontinence, nocturia and voiding frequency, as defined by the International Continence Society, referring to the previous four weeks.
  Overactive Bladder Questionnaire_V8 assessing severity of overactive bladder symptoms will be used. This scale includes items on urgency, incontinence, nocturia and voiding frequency, as defined by the International Continence Society. The final score is the sum of the partial scores obtained for each of the eight questions, ranging from 0 to 40.

SECONDARY OUTCOMES:
Urgency complaint assessed with the Perception of Intensity of Urgency Scale | Change from baseline urgency complaints at 6 weeks
  The patient's Perception of Intensity of Urgency Scale assessing urgency complaints will be used. This scale is scored on 0 and 4 points (the best score is '0' and the worst score is '4') based on urgency complaints. Higher scores indicate more severe urgency complaints.
Daily urinary frequency measured with voiding diary | Change from baseline the average daily urinary frequency at 6 weeks
  Patients will be also instructed to keep voiding diary for three days. In this diary, the average daily urinary frequency will be recorded.
The number of nocturia measured with voiding diary | Change from baseline the average number of nocturia at 6 weeks
  Patients will be also instructed to keep voiding diary for three days. In this diary, the average number of nocturia will be recorded.
The number of urinary incontinence measured with voiding diary | Change from baseline the average number of urinary incontinence at 6 weeks
  Patients will be also instructed to keep voiding diary for three days. In this diary, the average number of urinary incontinence will be recorded.
pelvic floor muscle strength measured with Modified Oxford Grading scale | Change from baseline pelvic floor muscle strength at 6 weeks
  The modified Oxford Grading Scale quantifies pelvic floor muscle strength as: 0, no contraction; 1, flicker; 2, weak; 3, moderate; 4, good; and 5, strong.
quality of life assessed with King's Health Questionnaire (KHQ) | Change from baseline quality of life at 6 weeks
  King's Health Questionnaire assessing quality of life related to urinary problems will be used. This questionnaire consists of two parts and 32 items. The first part (21 items) contains two single-item questions that address General Health Perception and Incontinence Impact and the following seven multi-item domains: Role, Physical, and Social Limitations, Limitations in Personal Relationship, Emotional Problems, Sleep and Energy Disturbances associated with UI, and Severity Measures for UI. The second part has an 11-item Symptom Severity Scale (SSS) that assesses the presence and severity of urinary symptoms. While the entire SSS is scored from 0 (best) to 30 (worst), the minimum possible score is 0 (best health) and the maximum possible score is 100 (worst health) for all other KHQ domains.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda TOPRAK CELENAY, Principal Investigator — Ankara Yildirim Beyazıt University; Zehra Korkut, Study Chair — KTO Karatay University; Kemal Oskay, Study Chair — Ankara Gazi Mustafa Kemal Hospital
Locations (1):
- Ankara Gazi Mustafa Kemal Hospital, Ankara, Turkey (Türkiye)